CLINICAL TRIAL: NCT07374211
Title: Effect of Esketamine on Perioperative Negative Emotions in Breast Cancer Surgery Patients With Severe Depression: A Randomized Controlled Trial
Brief Title: Effect of Esketamine on Perioperative Negative Emotions in Breast Cancer Surgery Patients With Severe Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PLAGH-RCT-Esket-SBreastCancer
Record Dates: First submitted 2026-01-18; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Depression; Anxiety; S-ketamine; Breast Cancer
MeSH Terms: conditions — Depression; Anxiety Disorders; Breast Neoplasms | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine group (Experimental): Patients who undergo general anesthesia using esketamine.
  Interventions: Drug: Esketamine 0.3mg/kg
- Control group (Placebo Comparator): Patients who undergo general anesthesia without esketamine
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Esketamine 0.3mg/kg — A single intravenous bolus of 0.3 mg/kg of esketamine is administered during anesthesia induction, and the infusion is completed over 40 minutes.
  Arms: Esketamine group
Drug: normal saline — Receiving the same volume of normal saline during induction of anesthesia.
  Arms: Control group

SUMMARY:
This project employs a prospective, randomized, controlled, blinded, dual-center study design to investigate the effects of intraoperative esketamine on perioperative anxiety and depression symptoms in patients with severe depression undergoing breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Scheduled to undergo elective breast cancer resection surgery.
3. American Society of Anesthesiologists (ASA) physical status classification of I-III.
4. Clearly understand and voluntarily agree to participate in the study, and sign the informed consent form.
5. Female patients with severe depressive symptoms (defined as a Hospital Anxiety and Depression Scale-Depression subscale score of ≥15)
6. Anticipated anesthesia duration greater than 90 minutes.

Exclusion Criteria:

1. Patients with significant preoperative abnormalities in cardiac, pulmonary, hepatic, or renal function, or coagulation disorders .
2. Patients taking antipsychotics, antidepressants, or glucocorticoids, or with a history of alcohol abuse or illicit drug use .
3. Patients with an MMSE score <18, dementia, intellectual disability, or those unable to communicate (e.g., coma, severe dementia, hearing or language impairment) .
4. Patients with a history of psychiatric or neurological disorders (e.g., schizophrenia, epilepsy, Parkinson's disease, or severe myasthenia gravis) .
5. Patients with poorly controlled or untreated hypertension (≥180/110 mmHg) .
6. Patients with elevated intracranial or intraocular pressure.
7. Patients with untreated or inadequately treated hyperthyroidism .
8. Patients with a known allergy to the drugs involved in this study .
9. Patients unable to complete the assessment scales required by this study.
10. Patients who are currently participating in other clinical trials

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2026-01-18 (Estimated); Primary Completion 2026-01-18 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative anxiety and depreession | Preoperative day 1, postoperative day 3 ,day 7 and day 30
  The primary outcomes were depression and anxiety, which were assessed using the Hospital Anxiety and Depression Scale . Perioperative anxiety was measured using the Hospital Anxiety and Depression Scale-Anxiety subscale, a standardized self-report instrument consisting of 7 items. Patients with a HADS-A score of 8 or more were considered to be experiencing anxiety, with a score of 8 to 10 indicating mild anxiety, 11 to 14 indicating moderate anxiety, and 15 to 21 indicating severe anxiety. Perioperative depression was measured using the Hospital Anxiety and Depression Scale-Depression subscale. Patients with a HADS-D score of 8 or more were considered to be experiencing depression, with a score of 8 to 10 indicating mild depression, 11 to 14 indicating moderate depression, and 15 to 21 indicating severe depression.

SECONDARY OUTCOMES:
Postoperative Sleep Quality | Preoperative day 1, postoperative day 3 ,day 7 and day 30
  Postoperative sleep quality was assessed using the Insomnia Severity Index (ISI). The ISI is a simple tool used to screen for insomnia and consists of 7 items to assess the nature and symptoms of the subject; sleep disorder on a 5-point Likert scale, with each item scored from 0 to 4 and the total score ranging from 0 to 28, with higher scores indicating greater severity of insomnia. The sum of the scores with 0-7 indicating insomnia without clinical significance, 8-14 indicating subclinical insomnia, 15-21 indicating clinical insomnia (moderate), 22-28 indicating 'clinical insomnia (moderate), and 22-28 indicating clinical insomnia (moderate). A score of 8 to 14 indicates subclinical insomnia, a score of 15 to 21 indicates clinical insomnia (moderate), and a score of 22 to 28 indicates clinical insomnia (severe).
Delirium | Within 7 days after surgery
  Delirium was assessed using a combination of the 3-Minute Diagnostic Interview for CAM (3D-CAM) and the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Patients in the general ward were assessed using the 3D-CAM, while patients in the intensive care unit were assessed using the CAM-ICU. Delirium consists of four main features: acute altered mental status or fluctuating level of consciousness, inattention, disorganized thinking, and altered level of consciousness. Patients were diagnosed with postoperative delirium if both the first and second features were present, and either the third or fourth feature was also present.
PONV | Within 2 days after extubation
  Postoperative nausea and vomiting (PONV) were assessed using a visual analogue scale (VAS). This scale consists of a 10-centimeter straight line, with 0 indicating no nausea and vomiting, and 10 indicating the most extreme level of nausea and vomiting that can be endured. The severity of PONV is categorized as follows: mild (1 to 4), moderate (5 to 6), and severe (7 to 10).
Postoperative Recovery Quality | Postoperative day 3 ,day 7 and day 30
  Postoperative quality of recovery was evaluated using the Chinese version of the Quality of Recovery-15 (QoR-15) score. This assessment tool comprises 15 items, each scored on a 10-point scale. The total score ranges from 0 to 150, with 0 indicating poor recovery and 150 signifying an excellent quality of recovery
Postoperative Pain | Postoperative day 3 ,day 7 and day 30
  Assessment was conducted using the Numerical Rating Scale (NRS) for pain, which ranges from 0 to 10. On this scale, a score of 0 represents the absence of pain, while a score of 10 represents the most severe pain.
Postoperative Quality of Life | postoperative day 3 ,day 7 and day 30
  Postoperative quality of life was assessed using the EuroQol 5-Dimension questionnaire (EQ-5D). This instrument evaluates five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For the descriptive system, each dimension is typically rated using a three-level scale (no problems, some problems, extreme problems) or a five-level scale (no problems, slight problems, moderate problems, severe problems, extreme problems).The responses are combined to form a 5-digit health state profile (e.g., 11111 for no problems in any dimension). This profile is then converted into a single summary number called the EQ-5D index score, using a country-specific value set. The theoretical range of the index score is approximately from -0.594 (worst imaginable health state, considered worse than death) to 1.0 (perfect health), with 0 representing a health state equivalent to death. Therefore, a higher EQ-5D index score indicates a better quality of life.

OTHER OUTCOMES:
Intraoperative blood pressure | During the surgery
Intraoperatively heart rate | During the surgery
Perioperative inflammatory factor (IL-6) | perioperatively
Perioperative brain injury-related factor (S100β) | perioperatively
Perioperative brain-derived neurotrophic factor (BDNF) | perioperatively
Perioperative acetylcholine (Ach) | perioperatively
Perioperative norepinephrine (NE) | perioperatively

IPD SHARING:
Plan to Share IPD: No